CLINICAL TRIAL: NCT01607294
Title: A Placebo-Controlled, Randomized, Double-Blind, Parallel Group, Single Center Study to Evaluate the Efficacy and Safety of ETC 1002 in Subjects With Type 2 Diabetes
Brief Title: A Single Center Study to Evaluate the Efficacy and Safety of ETC 1002 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Esperion Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1002-005
Record Dates: First submitted 2012-04-26; First posted 2012-05-30 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Hyperlipidemia; Type 2 Diabetes
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus, Type 2 | interventions — 8-hydroxy-2,2,14,14-tetramethylpentadecanedioic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ETC-1002 (Experimental): ETC-1002 daily Weeks 1-2, 80 mg/day; Weeks 3-4, 120 mg/day
  Interventions: Drug: ETC-1002
- Placebo (Placebo Comparator): Placebo daily 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ETC-1002 — ETC-1002 Daily for 4 weeks
  Arms: ETC-1002
Drug: Placebo — Placebo Daily for 4 weeks
  Arms: Placebo

SUMMARY:
This Phase 2 study will asses the LDL-C lowering efficacy of ETC-1002 versus placebo in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes meeting all of the following:
* Minimum 6 month history of diabetes prior to screening visit;
* Fasting C-peptide ≥ 0.8 ng/mL at screening visit;
* HbA1C at screening visit 7-10%;
* Fasting glucose from 140-270 mg/dL on Day -7 following washout of all glucose regulating drugs and supplements.
* BMI at screening visit from 25-35 kg/m2;
* LDL-C at screening ≥ 100 mg/dL

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
assess the LDL-C lowering efficacy of ETC-1002 versus placebo in subjects with type 2 diabetes | 4 weeks
  evaluate the change in LDL-C from baseline to various time points

SECONDARY OUTCOMES:
assess the effect of ETC-1002 versus placebo on glycemic parameters including fasting plasma and postprandial glucose and insulin | 4 weeks
  evaluate the change in glucose and insulin from baseline to various time points
assess the effect of ETC-1002 versus placebo on measures of insulin sensitivity in subjects with type 2 diabetes | 4 weeks
  evaluate the change in HOMA-IR from baseline to various time points
assess safety using adverse event reports, physical exams, vital signs, ECGs and clinical laboratory parameters | 4 weeks
  evaluate any changes in safety parameters during the course of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Miramar, Florida, United States

REFERENCES:
- [Derived] Gutierrez MJ, Rosenberg NL, Macdougall DE, Hanselman JC, Margulies JR, Strange P, Milad MA, McBride SJ, Newton RS. Efficacy and safety of ETC-1002, a novel investigational low-density lipoprotein-cholesterol-lowering therapy for the treatment of patients with hypercholesterolemia and type 2 diabetes mellitus. Arterioscler Thromb Vasc Biol. 2014 Mar;34(3):676-83. doi: 10.1161/ATVBAHA.113.302677. Epub 2014 Jan 2. PMID 24385236